CLINICAL TRIAL: NCT04712643
Title: A Phase III, Open-Label, Randomized Study of On-Demand TACE Combined With Atezolizumab Plus Bevacizumab (Atezo/Bev) or On-Demand TACE Alone in Patients With Untreated Heaptocellular Carcionma
Brief Title: A Study of TACE Combined With Atezolizumab Plus Bevacizumab or TACE Alone in Patients With Untreated Heaptocellular Carcionma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML42612
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: atezolizumab + bevacizumab + TACE (Experimental): Participants will receive atezolizumab plus bevacizumab on Day 1 of a 21-Day cycle, after every on-demand transarterial chemoembolization procedure.
  Interventions: Drug: Atezolizumab; Drug: Becavizumab; Device: Transarterial chemoembolization (TACE)
- Arm B: TACE alone (Active Comparator): Participants will receive on-demand transarterial chemoembolization.
  Interventions: Device: Transarterial chemoembolization (TACE)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until participant experience loss of clinical benefit as evaluated by the investigator or unacceptable toxicity or withdrawal of informed consent.
  Other Names: Tecentriq
  Arms: Arm A: atezolizumab + bevacizumab + TACE
Drug: Becavizumab — Bevacizumab will be administered by IV infusion at a fixed dose of 15 mg/kg on Day 1 of each 21-day Cycle.
  Other Names: Avastin
  Arms: Arm A: atezolizumab + bevacizumab + TACE
Device: Transarterial chemoembolization (TACE) — TACE will be performed by clinical demand.

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab plus bevacizumab combined with on-demand TACE compared to on-demand TACE alone in participants with hepatocellular carcinoma who are at high risk of poorer outcome following TACE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC by histology/ cytology or clinical criteria
* Eligible for TACE treatment
* No prior systemic therapy for HCC, especially immunotherapy
* No prior locoregional therapy to the target lesion(s)
* At least one measurable untreated lesion
* ECOG Performance Status of 0-1
* Child-Pugh class A

Exclusion Criteria:

* Evidence of Vp3/4 and hepatic vein tumor thrombus (HVTT)
* Evidence of extrahepatic spread (EHS)
* Being a candidate for curative treatments
* Any condition representing a contraindication to TACE as determined by the investigators
* Active or history of autoimmune disease or immune deficiency
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
TACE Progression-Free Survival (TACE PFS) as Determined by Investigator | Randomization to untreatable progression or TACE failure/refractoriness or death (up to approximately 46 months)
  TACE PFS is defined as the time from randomization to untreatable progression or TACE failure/refractoriness or any cause of death, whichever occurs first, as determined by the investigator (INV).
Overall Survival (OS) | Randomization to death from any cause (up to approximately 94 months)
  Overall survival (OS) after enrollment is defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Time to Untreatable (unTACEable) Progression (TTUP) as Determined by Investigator | Randomization to untreatable (unTACEable) progression (up to approximately 46 months)
  INV-assessed TTUP is defined as time from randomization to untreatable (unTACEable) progression, as determined by investigator.
Time to Progression (TTP) as Determined by Investigator | Randomization to unTACEable progression or TACE failure/refractoriness (up to approximately 46 months)
  INV-assessed TTP is defined as the time from randomization to unTACEable progression or TACE failure/refractoriness (as defined above), as determined by investigator.
Time to Extrahepatic Spread (EHS) as Determined by Investigator | Randomization to first evidence of EHS (up to approximately 46 months)
  INV-assessed time to EHS is defined as the time from randomization to the first evidence of EHS, as determined by investigator.
Objective Response Rate (ORR), as Determined by Investigator | Randomization up to approximately 46 months
  Objective response (OR) is defined as a complete or partial response, as determined by investigator.
Duration of Responses (DOR) as Determined by Investigator | First occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first)(up to approximately 46 months)
  INV-assessed DOR is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by INV.
Progression Free Survival (PFS) | Randomization to first occurrence of disease progression or death from any cause (whichever occurs first)(up to approximately 94 monthsJ)
  Progression free survival (PFS) is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Time to Deterioration (TTD) | Randomization to first deterioration (up to approximately 94 months)
  TTD is defined as the time from randomization to first deterioration in the patient-reported GHS/QoL, physical function, or role function scales of the EORTC QLQ-C30, maintained for two consecutive assessments, or one assessment followed by death from any cause within 3 weeks.
Percentage of Participants With Adverse Events | Baseline up to approximately 94 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- China (30):
  - Anhui Provincial Hospital, Anhui
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing You An Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Southwest Hospital , Third Military Medical University, Chongqing
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Fujian Cancer Hospital, Fuzhou
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan Unvierstiy, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xi'an Inernational Medical Center Hospital, Xi'an
  - Henan Cancer Hospital, Zhengzhou
  - Zhuhai People's Hospital, Zhuhai
- Japan (10):
  - Aichi Cancer Center, Aichi
  - Chiba University Hospital, Chiba
  - Kurume University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Yokohama City University Medical Center, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - The University of Osaka Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Toranomon Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing